CLINICAL TRIAL: NCT06451523
Title: Effects of "Alliance180 Program" on Psychological and Physical Well-Being
Brief Title: Effects of "Alliance180 Program" on Well-Being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: ALLIANCE180, INC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-2072
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Trauma and Stressor Related Disorders
Keywords: Anxiety Depression; Autonomic Reactivity; Polyvagal Theory
MeSH Terms: conditions — Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: All participants will follow the same procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alliance180 Program (Experimental): Participants will attend the 3-day Alliance180 Program.
  Interventions: Other: Alliance180 Program

INTERVENTIONS:
Other: Alliance180 Program — The Alliance180 Program promotes feelings of neuropsychological safety and trust in the context of a 3-day program, which includes the transformative equine experience.

SUMMARY:
The goal of this clinical trial is to evaluate the effects of the Alliance180 Program on physical and psychological well-being on adults who are/were US Veterans, First Responders and/or Front Line Healthcare Workers.

The study aims are:

* Aim #1: to evaluate the effect of the Alliance180 Program on physical and psychological well-being in adults who are/were US Veterans, First Responders and/or Front Line Healthcare Workers;
* Aim #2: to evaluate the relationship between between feelings of safety and well-being, autonomic functioning, and mental health indices (depression, anxiety, trauma response) before and after the intervention.

Participants will be asked to complete self-report measures of feelings of safety and well-being, autonomic functioning, and mental health indices (depression, anxiety, trauma response) before participating in the Alliance180 Program (i.e., baseline research session) and 1 week, 1 month, 3 months and 6 months after completing the Alliance180 Program. Demographic information will be documented during the baseline research session.

DETAILED DESCRIPTION:
All data collection will occur remotely using REDCap (via University of North Carolina, Chapel Hill). As this is a single-arm, feasibility/pilot study, all participants will follow the same protocol.

1. Baseline Research Session: self-report completion of demographic information, perception of safety (Neuroception of Psychological Safety, NPSS) and trauma experience (Posttraumatic Stress Disorder Checklist DSM-5, PCL-5), autonomic reactivity (Body Perception Questionnaire, BPQ), anxiety/depression (Hospital Anxiety and Depression Scale, HADS), and perception of events and goals related to purpose in life (Purpose in Life Scale).
2. Participate in the 3-day Alliance180 Program (intervention), which includes the Transformative Equine Experience.
3. Post-intervention Research Sessions: 1 week, 1 month, 3 months and 6 months after completing the Alliance180 Program, self-report completion of perception of safety and trauma experience (NPSS, PCL-5), autonomic reactivity (BPQ), anxiety/depression (HADS) and purpose of events and goals related to purpose in life (Purpose in Life Scale).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Enrollment in an upcoming "Alliance180 Program". (Enrollment is limited to adults who currently or formerly serve as US Veterans, First Responders and/or Front Line Healthcare Workers and are currently experiencing symptoms related to trauma exposure)

Exclusion Criteria:

- Individuals who have previously completed the "Alliance180 Program"

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Anxiety Subscale of the Hospital Anxiety and Depression Scale | Baseline, 1 month
  The Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of anxiety over the prior week. The anxiety subscale ranges from 0 to 21, with higher scores indicating higher anxiety complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Depression Subscale of the Hospital Anxiety and Depression Scale | Baseline, 1 month
  The Depression Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of depression over the prior week. The depression subscale ranges from 0 to 21, with higher scores indicating higher depression complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.

SECONDARY OUTCOMES:
Change in the Body Perception Questionnaire | Baseline, 1 month
  Body Perception Questionnaire (BPQ) is a self-report questionnaire, which includes a 20-item subscale for Autonomic Nervous System Reactivity. Only the Autonomic Nervous System Reactivity subscale will be administered. Raw scores range from 0-100, with higher scores indicating greater level of symptoms associated with autonomic activity (poorer outcome). Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Neuroception of Psychological Safety Scale | Baseline, 1 month
  Neuroception of Psychological Safety Scale (NPSS) is a self-report questionnaire, which contains 29-items. Raw scores range from 29-145, with higher scores indicating stronger feelings of psychological safety. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Posttraumatic Stress Disorder Checklist (DSM-5) | Baseline, 1 month
  Posttraumatic Stress Disorder Checklist (DSM-5) (PCL-5) is a self-report questionnaire, which contains 20-items. Raw scores range from 0-80, with higher scores indicating more symptoms of PTSD. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Purpose in Life Questionnaire | Baseline, 1 month
  Purpose in Life Questionnaire is a self-report questionnaire, which contains 12-items. Raw scores range from 0-60, with higher scores indicating a greater sense of purpose in life. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Anxiety Subscale of the Hospital Anxiety and Depression Scale | Baseline, 6 months
  The Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of anxiety over the prior week. The anxiety subscale ranges from 0 to 21, with higher scores indicating higher anxiety complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Depression Subscale of the Hospital Anxiety and Depression Scale | Baseline, 6 months
  The Depression Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of depression over the prior week. The depression subscale ranges from 0 to 21, with higher scores indicating higher depression complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Body Perception Questionnaire | Baseline, 6 months
  Body Perception Questionnaire (BPQ) is a self-report questionnaire, which includes a 20-item subscale for Autonomic Nervous System Reactivity. Only the Autonomic Nervous System Reactivity subscale will be administered. Raw scores range from 0-100, with higher scores indicating greater level of symptoms associated with autonomic activity (poorer outcome). Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Neuroception of Psychological Safety Scale | Baseline, 6 months
  Neuroception of Psychological Safety Scale (NPSS) is a self-report questionnaire, which contains 29-items. Raw scores range from 29-145, with higher scores indicating stronger feelings of psychological safety. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Posttraumatic Stress Disorder Checklist (DSM-5) | Baseline, 6 months
  Posttraumatic Stress Disorder Checklist (DSM-5) (PCL-5) is a self-report questionnaire, which contains 20-items. Raw scores range from 0-80, with higher scores indicating more symptoms of PTSD. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Change in the Purpose in Life Questionnaire | Baseline, 6 months
  Purpose in Life Questionnaire is a self-report questionnaire, which contains 12-items. Raw scores range from 0-60, with higher scores indicating a greater sense of purpose in life. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Keri J Heilman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Alliance180, Saratoga Springs, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina, Chapel Hill (UNC).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 and continuing for 36 months after publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina, Chapel Hill (UNC).